CLINICAL TRIAL: NCT01554072
Title: Home-based Pulmonary Rehabilitation in COPD
Brief Title: Home-based in Chronic Obstructive Pulmonary Disease
Acronym: HBCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fernanda Dultra Dias, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 384767; pulmonary rehabilitation (Registry Identifier: Home-based pulmonary rehabilitation in COPD)
Record Dates: First submitted 2012-01-17; First posted 2012-03-14 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: home-based; pulmonary rehabilitation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive a booklet of exercises, besides containing an explanation of his illness and the importance of exercise in their quality of life, an exercise routine physical to be held three times a week for two consecutive months. Patients will be instructed individually on each exercise, performing with supervisor that there be no doubt about execution, thereby minimizing any possible mistake in practice at home. For each day of the year ended data should be recorded in a daily monitoring. At the end of two months of the PR program semi-home patients will be subject to review so that all tests should be applied again.
  Interventions: Other: Home based pulmonary rehabilitation with exercise
- exercise (Active Comparator): Patients will receive a booklet of exercises, besides containing an explanation of his illness and the importance of exercise in their quality of life, an exercise routine physical to be held three times a week for two consecutive months. For each day of the year ended data should be recorded in a daily monitoring. Is also scheduled a visit to the laboratory biweekly in which patients demonstrate their exercise routine program RP semi-home settings for any load, postural corrections and execution of physical exercise, should be refocused. At the end of two months of the PR program semi-home patients will be subject to review so that all tests should be applied again.
  Interventions: Other: Home based pulmonary rehabilitation with exercise

INTERVENTIONS:
Other: Home based pulmonary rehabilitation with exercise — After each group will receive the randomization their booklets containing the exercise routine that should be performed at home., to be held three times a week for two consecutive months. Is also scheduled a visit to the laboratory biweekly Respiratory Functional Assessment in which patients demonstrate their exercise routine program RP semi-home settings for any load, postural corrections and execution of physical exercise, should be refocused.

SUMMARY:
Pulmonary rehabilitation consists of a multidisciplinary program of care for patients with chronic respiratory disease, which currently encompasses numerous features and physical training methods aimed at maintaining stability clinic for people with Chronic Obstructive Pulmonary Disease (COPD), especially in patients who, even with optimized clinical treatment, continue their decline and symptomatic physical functions and 8 so that these social. goals are achieved the patient with COPD should integrate into a program of RP assiduous and with accompanying several times per week, for several months, which for a number of factors is not always possible. For this reason, it is the research of methodology of RP that hold their effectiveness, but with greater flexibility and viability to people with COPD. On this basis, this study aims to investigate the effectiveness of a program of RP semi-domiciliar in which the patient suffering from COPD can receive guidance and training in person, to develop it partially in own domicile.

DETAILED DESCRIPTION:
The protocol of the experimental procedure will begin with the explanation of the purpose, risks and benefits of the study volunteers to patients with COPD. Subsequently, based on an evaluation form, will collect data on the past history and current disease and performed a general physical examination. Then the patients will respond to two questionnaires. The first will research the Medical Council (MRC) 13, which is a dyspnea scale to categorize in terms of disability, patients with COPD. The second questionnaire will be the Airway Questionnaire 20 (AQ20) 14 specific for obstructive pulmonary disease, which is validated for the local language and highly reliable for the evaluation of patients with COPD, containing 20 questions related to respiratory health to evaluate the quality of life. Subsequently, the same day, the patients carry out the following tests: spirometry, respiratory muscle strength, respiratory muscle endurance, assessment of training load of the upper and shuttle test and bioimpedance

ELIGIBILITY:
Inclusion Criteria:

* will be included patients of both sexes,
* over 40 years and diagnosis of COPD according to criteria of ATS, GOLD and II Brazilian Consensus of COPD.
* must be medically stable,
* without having presented the framework of exacerbation of disease over the past 30 days and,
* must have agreed to participate in this study which, after being presented and explained to patients, this accepted should be confirmed by Subscription Term of free and informed consent, pursuant to resolution 96 of 1996 of MS.

Exclusion Criteria:

* will be excluded from the study patients with serious comorbidity,
* orthopedic diseases such as heart defects in upper and lower limbs,
* sequelae of motor neurological disorders or impaired that may interfere with the ability to carry out physical exercise,
* uncontrolled hypertension,
* lung diseases and
* those who do not grant support to participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of functional capacity and quality of life after Home-based rehab | After two months of treatment
  Observe the effectiveness of home rehabilitation on functional capacity and quality of life among the placebo group and intervention as well as pre and post assessment patient care intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Dias, Principal Investigator — University of Nove de Julho
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Dias FD, Sampaio LM, da Silva GA, Gomes EL, do Nascimento ES, Alves VL, Stirbulov R, Costa D. Home-based pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a randomized clinical trial. Int J Chron Obstruct Pulmon Dis. 2013;8:537-44. doi: 10.2147/COPD.S50213. Epub 2013 Nov 5. PMID 24235824